CLINICAL TRIAL: NCT07297563
Title: A Randomized, Open-label Study To Compare The Efficacy And Safety Of Anti-CD38 Monoclonal Antibody Versus Rituximab in ITP Patients Who Failed or Relapsed After Glucocorticoid Therapy
Brief Title: Anti-CD38 Monoclonal Antibody Versus Rituximab in the Management of Primary Immune Thrombocytopenia (ITP)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2023067
Record Dates: First submitted 2025-11-21; First posted 2025-12-22 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Immune Thrombocytopenia; Treatment
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Rituximab; daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rituximab (Active Comparator): Rituximab (375mg/m2) was given once.
  Interventions: Drug: Rituximab
- Daratumumab（Anti-CD38 Monoclonal Antibody ） (Experimental): Daratumumab（anti-CD38 monoclonal antibody ）(16mg/kg) was given once a week for eight times
  Interventions: Drug: Daratumumab

INTERVENTIONS:
Drug: Rituximab — All subjects were randomly assigned to group A (active comparator) and group B (experimental). For subjects in group A (active comparator) , rituximab (375mg/m2) was given once.
  Arms: rituximab
Drug: Daratumumab — All subjects were randomly assigned to group A (active comparator) and group B (experimental). For subjects in group B (experimental), Daratumumab (anti-CD38 monoclonal antibody ) (16mg/kg) was given once a week for eight times.
  Arms: Daratumumab（Anti-CD38 Monoclonal Antibody ）

SUMMARY:
This randomized, open-label study aim to compare the efficacy and safety of Daratumumab (anti-CD38 monoclonal antibody) with rituximab in ITP patients.This study will be conducted in ITP patients who had not responded to or had relapsed after previous glucocorticoid treatment.

DETAILED DESCRIPTION:
Immune thrombocytopenia (ITP) is an organ-specific autoimmune disease, which is characterized by decreased platelet count and skin and mucosal bleeding. ITP is a kind of disease with increased platelet destruction and impaired platelet production caused by autoimmunity. Conventional treatment of adult ITP includes first-line glucocorticoid and immunoglobulin therapy, second line TPO and TPO receptor agonist, splenectomy and other immunosuppressive treatments (such as rituximab, vincristine, azathioprine, etc.). ITP is one of the most common hemorrhagic diseases. At present, the treatment response of ITP is not good, and a considerable number of patients need drug maintenance treatment, which seriously affects the quality of life of patients and increases the economic burden of patients. Therefore, there is still a lack of effective treatment for adult ITP, especially for recurrent and refractory ITP patients, which is one of the problems that have attracted more attention and need to be solved urgently.

The main pathogenesis of ITP is the loss of platelet autoantigen immune tolerance, which leads to abnormal activation of humoral and cellular immunity. It is characterized by antibody mediated platelet destruction and insufficient platelet production by megakaryocytes. The residual long-term autoreactive plasma cells may be a source of therapeutic resistance to autoimmune cytopenia. Antiplatelet specific plasma cells have been detected in the spleen of patients with rituximab refractory ITP. Therefore, the strategy of simply eliminating B cells may not work, because LLPC will continue to produce pathogenic antibodies. In view of this, anti-CD38 monoclonal antibody can eliminate LLPC, thereby profoundly reducing the production of pathogenic antibodies and achieving good efficacy. Some patients have been treated with this Daratumumab (anti-CD38 monoclonal antibody) in the past, with good efficacy and safety. Therefore, the investigator planned to conduct a clinical study to evaluate the safety and efficacy of Daratumumab (anti-CD38 monoclonal antibody) versus rituximab in relapsed adult patients with primary immune thrombocytopenia, in order to provide more treatment options for patients with ITP.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years, male or female.
* Before enrollment, the subjects have been clinically diagnosed with primary immune thrombocytopenia for no less than three months according to the American Society of Hematology guidelines 2011 Evidence-Based Practice Guideline (Neunert et al. 2011) or the International Consensus Report for the Investigation and Management of Primary Immune Thrombocytopenia (Provan et al. 2010), as applicable locally.
* Patients have failed glucocorticoid therapy (either due to inefficacy, efficacy could not be maintained, or relapse). Patients were required to have a response history (PLT≥50×10^9/L) to standard first-line treatment of ITP (glucocorticoid and/or intravenous immunoglobulin).
* Subjects with a platelet count of <30×10^9/L within the 24 hours prior to the first dose of the study drug; The mean platelet count of at least two separate assessments (at least 1 week apart) <30×10^9/L during the screening visit, and no platelet count > 35×10^9/L.
* ECOG performance status score of ≤2.
* Enrollment of subjects receiving maintenance therapy with a stable dosage is permitted, including glucocorticoids (≤0.5 mg/kg of prednisone or equivalent) or TPO receptor agonists. However, at the time of enrollment, subjects are restricted to using only one concomitant medication with a stable dose, and the concomitant medication must have been stable for a minimum of 4 weeks prior to the initial infusion of the study drug.
* For fertile female patients, a negative pregnancy test result is required. Fertile female and male patients must use effective contraception separately during the study and for 4 or 6 months after the cessation of study drug treatment.
* Subjects comprehensively understand and can adhere to the study protocol requirements and willingly signed the informed consent form.

Exclusion Criteria:

* Subjects with a history of using CD20 monoclonal antibody or CD38 monoclonal antibody.
* Subjects who are diagnosed with autoimmune hemolytic anemia or various secondary thrombocytopenic disorders.
* Subjects with history of any thrombotic or embolic events or extensive and severe bleeding, such as hemoptysis, major upper gastrointestinal bleeding, intracranial hemorrhage, or the presence of sepsis or other irregular bleeding within the 12 months preceding the initiation of the first dose of study drug.
* Subjects who have participated in any other investigational drug studies (including vaccine studies) or been exposed to other investigational drugs within the first 4 weeks or 5 half-lives (whichever was longer) prior to the first dose of study drug.
* Subjects who have used anticoagulants or any agents with antiplatelet effects, such as aspirin, within 3 weeks prior to the first dose of study drug.
* Subjects who have received emergency treatment for ITP (e.g., methylprednisolone, platelet transfusion, intravenous immunoglobulin infusion, or thrombopoietin receptor agonist therapy) within 2 weeks prior to the first dose of study drug.
* Subjects who have been treated with medications including azathioprine, danazol, dapsone, cyclosporine A, tacrolimus, and sirolimus within 4 weeks prior to the first dose of study drug. Subjects who have receive medications including cyclophosphamide and vindesine within 6 months prior to the first dose of study drug.
* Subjects who have undergone splenectomy within 6 months prior to the first dose of study drug.
* Subjects who have received live vaccines within 4 weeks prior to the first dose of study drug, or plan to receive any live vaccines during the course of the study.
* Subjects who are diagnosed with Myelodysplastic syndromes (MDS); Subjects with a with a history of malignancy within the 5 years prior to screening (excluding completely cured in situ cervical cancer and non-metastatic skin squamous cell carcinoma or basal cell carcinoma).
* Subjects who have undergone allogeneic stem cell transplantation or organ transplantation.
* Subjects with a clinically significant medical history, as perceived by investigators, that will pose risks to subjects' safety during the study or potentially affect the safety or efficacy analyses, includes major clinical histories such as circulatory system abnormalities, endocrine system abnormalities, nervous system diseases, blood system diseases, immune system diseases, mental diseases and metabolic abnormalities and so on. e.g., subjects with acute myocardial infarction, unstable angina pectoris, or severe arrhythmias (multifocal ventricular premature contractions, ventricular tachycardia, or ventricular fibrillation) within the 6 months before screening ; New York Heart Association (NYHA) class III-IV heart failure; subjects who were known to have had moderate or severe persistent asthma or chronic obstructive pulmonary disease within the 5 years prior to screening, or whose condition was currently poorly controlled;
* Subjects with a history of severe recurrent or chronic infections, or acute infections requiring systemic treatment with antibiotics, antiviral drugs, antiparasitic drugs, anti-amoebic drugs, or antifungal drugs within 4 weeks prior to the first dose and during the screening period, or superficial skin infections requiring systemic treatment within one week prior to the first dose of study drug. Notably, after the resolution of the infection, the subject may be re-screened.
* Subjects with a history of known or suspected immunosuppression, including invasive opportunistic infections such as histoplasmosis, listeriosis, coccidioidomycosis, pneumocystis pneumonia, and aspergillosis, even if the infection has resolved; or unusually frequent, recurrent, or prolonged infections (as judged by the investigator).
* Significant laboratory abnormalities during screening included:

  1. Alanine aminotransferase or aspartate aminotransferase greater than three times the upper limit of normal (ULN).
  2. Total bilirubin greater than 1.5 times the ULN (note: subjects diagnosed with Gilbert syndrome based on medical records should not be excluded based on this criterion).
  3. absolute neutrophil count < 1500/mm3.
  4. hemoglobin < 9g/dL.
  5. IgG < 500 mg/dL.
  6. lymphocyte count < 500/mm3.
  7. Creatinine clearance (CrCl) < 30 mL/min (i.e., CrCl ≥30 mL/min is allowed)
* Positive for HIV antibodies or syphilis antibodies.
* Subjects test positive for Hepatitis B surface antigen (HBsAg) or subjects test positive for hepatitis B core antibody and HBV-DNA (through polymerase chain reaction testing), or subjects test positive for hepatitis C virus antibody and HCV-RNA during the screening period. Subjects with positive hepatitis B core antibody but negative HBV-DNA can be enrolled, with HBV-DNA monitoring every 4 weeks.
* Pregnant or lactating women, or those intending to conceive or breastfeed during the study; and male partners intending to induce pregnancy during the study.
* Any other conditions unsuitable for participation in this study, as assessed by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-01-20 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Overall response rate at week 12 | 12 weeks
  Overall response rate was defined as proportion of subjects with a platelet count ≥ 30 × 10^9/L and at least twice the baseline platelet count without bleeding at week 12 after initial administration in absence of rescue therapy, and without having had dose increment of TPO-RA or corticosteroids during the study period.

SECONDARY OUTCOMES:
Complete response rate at week 12 | 12 weeks
  Complete response rate was defined as proportion of subjects with a platelet count ≥ 100 × 10^9/L without bleeding at week 12 after initial administration in absence of rescue therapy, and without having had dose increment of TPO-RA or corticosteroids during the study period.
Partial response rate at week 12 | 12 weeks
  Partial response rate was defined as proportion of subjects with a platelet count ≥30 to <100 × 10^9/L and at least twice the baseline platelet count without bleeding at week 12 after initial administration in absence of rescue therapy, and without having had dose increment of TPO-RA or corticosteroids during the study period.
Overall response rate at week24 | 6 months
  Overall response rate was defined as proportion of subjects with a platelet count ≥ 30 × 10^9/L and at least twice the baseline platelet count without bleeding at week24 after initial administration in absence of rescue therapy, and without having had dose increment of TPO-RA or corticosteroids during the study period.
Overall response rate at week52 | 12 months
  Overall response rate was defined as proportion of subjects with a platelet count ≥ 30 × 10^9/L and at least twice the baseline platelet count without bleeding at week52 after initial administration in absence of rescue therapy, and without having had dose increment of TPO-RA or corticosteroids during the study period.
Proportion of subjects with a platelet count≥ 30×10^9/L and at least two times of baseline platelet count, ≥ 50 × 10^9/L and ≥ 100 × 10^9/L at each visit | 12 months
  Proportion of subjects with a platelet count≥ 30×10^9/L and at least two times of baseline platelet count, ≥ 50 × 10^9/L and ≥ 100 × 10^9/L at each visit after administration
Duration from treatment initiation to platelet count ≥30×10^9/L and at least two times of baseline platelet count, platelet count ≥50×10^9/L, platelet count ≥100×10^9/L | 12 months
  Duration from treatment initiation to platelet count ≥30×10^9/L and at least two times of baseline platelet count, platelet count ≥50×10^9/L, platelet count ≥100×10^9/L
Proportion of subjects receiving emergency treatment | 12 weeks
  Proportion of subjects receiving emergency treatment within 12 weeks and throughout the clinical trial
Concomitant maintenance drug | 12 weeks
  Changes in concomitant maintenance therapy at week12 compared with that before the study.
Changes in world health organization (WHO) bleeding scale | 12 months
  Changes in world health organization (WHO) bleeding scale without emergency treatment. Changes of every subject in WHO bleeding score after treatment according to the reported World Health Organization's Bleeding Scale. The WHO Bleeding Scale is a measure of bleeding severity with the following grades: grade 0 = no bleeding, grade 1= petechiae, grade 2= mild blood loss, grade 3 = gross blood loss, and grade 4 = debilitating blood loss.
Adverse events assessment | 12 months
  Incidence, severity, and relationship of treatment emergent adverse events after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Academy of Medical Science and Blood Disease Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Researchers qualified can request the dataset, including de-identified individual subject data. Data may be requested from PI from 12 months 36 months after study completion.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 12 months to 36 months after study completion
Access Criteria: Upon request to PI